CLINICAL TRIAL: NCT00244842
Title: A Phase III, Randomized, Multicentre, Double-Blind, Placebo-Controlled Study of ISA247 in Plaque Psoriasis Patients
Brief Title: Randomized Placebo-controlled Study of ISA247 in Plaque Psoriasis
Acronym: SPIRIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISA04-03
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Psoriasis
Keywords: Randomized Controlled Trials; Immunosuppression; Adult; Chronic Disease; Dermatologic Agents; Female; Humans; Male; Middle Aged; Severity of Illness Index; Treatment Outcome; Quality of Life; Double-Blind Method
MeSH Terms: conditions — Psoriasis; Chronic Disease | interventions — voclosporin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo Comparator: 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Voclosporin 0.2 mg/kg po BID (Active Comparator): Voclosporin 0.2 mg/kg po BID
  Interventions: Drug: voclosporin
- Voclosporin 0.3 mg/kg po BID (Active Comparator): Voclosporin 0.3 mg/kg po BID
  Interventions: Drug: voclosporin
- Voclosporin 0.4 mg/kg po BID (Active Comparator): Voclosporin 0.4 mg/kg po BID
  Interventions: Drug: voclosporin

INTERVENTIONS:
Drug: voclosporin — voclosporin 0.2, 0.3, or 0.4 mg/kg po BID
  Arms: Voclosporin 0.2 mg/kg po BID; Voclosporin 0.3 mg/kg po BID; Voclosporin 0.4 mg/kg po BID
Drug: Placebo — Placebo
  Arms: Placebo Comparator: 1

SUMMARY:
The purpose of this study is to determine which dose of voclosporin is effective in the treatment of plaque psoriasis compared to placebo.

DETAILED DESCRIPTION:
Psoriasis is a chronic skin condition that can have a significant impact on patient's physical and mental well being. The most common form of psoriasis is plaque psoriasis. Targeted treatments in psoriasis have been reported recently, yet cyclosporine, a calcineurin inhibitor (CNi) remains one of the treatments which has the greatest efficacy. Voclosporin represents the possibility of a calcineurin inhibitor which is not only as efficacious as cyclosporine A, but also has an improved toxicity profile.

Comparison(s): Voclosporin at 3 dose levels (0.2, 0.3, and 0.4 mg/kg twice a day)compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Plaque psoriasis ≥ 6 months prior to screening.
* Diagnosis of stable, plaque psoriasis; i.e. psoriasis must not be spontaneously improving or worsening in the 4 weeks prior to the screening visit.
* Plaque psoriasis involving ≥10% of the body surface area (BSA) at screening and prior to randomization at the day 0 visit.
* PASI score ≥10 at screening and prior to randomization at the day 0 visit.
* Not pregnant or nursing or planning to become pregnant during the course of the study.
* Sexually active women of childbearing potential or less than 1 year post-menopausal and sexually active men who are not surgically sterile must use a reliable form of birth control during study treatment and for at least 3 months after the last dose of study drug. Surgically sterile females are not considered to be of childbearing potential. Reliable forms of birth control include oral or depot contraceptives, and double-barrier methods.
* Written informed consent prior to washout and screening procedures.
* Able to keep study appointments and cooperate with all study requirements, in the opinion of the investigator.

Exclusion Criteria:

* Has generalized erythrodermic, guttate, or pustular psoriasis.
* Have other dermatoses that would interfere with the evaluation of psoriasis, at the discretion of the investigator.
* A current malignancy or history of malignancy within 5 years or a history of lymphoma at any time. Subjects can be enrolled with a history of squamous or basal cell carcinoma that has been surgically excised or removed with curettage and electrodesiccation.
* Has current, uncontrolled bacterial, viral, or fungal infections that require intravenous antibiotics or antifungals or had had such infections within 60 days prior to screening.
* A history of streptococcal infection that required oral antibiotics within 30 days prior to screening.
* A known history of tuberculosis.
* Serologic evidence or known latent human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C (HCV) virus.
* Uncontrolled hypertension as defined by systolic blood pressure ≥150 mm Hg or diastolic blood pressure ≥ 90 mm Hg.
* MDRD GFR ≤ 60 ml/min.
* Variation between the screening and Visit 1 GFR ≥30%.
* Alanine transaminase, aspartate transaminase, or gamma-glutamyl transferase ≥ 3x upper limit of normal (ULN).
* White blood cell count ≤ 2.8 x 109/L.
* Triglycerides ≥ 3x ULN.
* Requires the following prohibited medications or treatments during the washout or treatment period: drugs potentiating the nephrotoxicity of voclosporin such as NSAID's or ACE inhibitors, drugs interfering with its pharmacokinetics; drugs considered to contribute to psoriasis flare; or, systemic and topical psoriasis medication (including psoralen/ultraviolet A light treatment) that may interfere with assessment of study drug efficacy.
* Has used any investigational drug or device within 28 days or 5 half lives (whichever is longer) prior to the screening visit.
* Has taken biological agent(s), except flu shots, tetanus shots, or boosters, within 3 months of the start of treatment. Biological agents include any virus, therapeutic serum, toxin, antitoxin, or analogous product applicable to the prevention, treatment, or cure of diseases or injuries of man.
* Previous exposure to voclosporin.
* A history of clinically defined allergy to cyclosporine or any of the constituents of the voclosporin formulation (vitamin E, medium chain triglyceride oil, Tween 40, ethanol).
* A history of alcoholism or drug addiction within 1 year prior to study entry.
* Weighs <45 kg (99 lbs) or > 140 kg (308 lbs).
* A history of disease, including mental/emotional disorder that would interfere with the subject's participation in the study, or that might cause the administration of ISA247 to pose a significant risk to the subject, in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2004-12; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research; Richard Langley, MD, FRCPC, Principal Investigator — Eastern Canada Cutaneous Research Associates Ltd.; Gilles Lauzon, PhD MD FRCPC, Principal Investigator — Western Canada Dermatology Institute; Kim Papp, MD, PhD, Principal Investigator — Probity Medical Research; Neil Shear, MD, Principal Investigator — Ventana Clinical Research Organization
Locations (25):
- Canada (25):
  - Isotechnika Investigational Site, Calgary, Alberta
  - Isotechnika Investigational Site', Edmonton, Alberta
  - Isotechnika Investigational Site, Edmonton, Alberta
  - Isotechnika Investigational Site, Vancouver, British Columbia
  - Isotechnika Investigational Site, Victoria, British Columbia
  - Isotechnika Investigational Site, Winnipeg, Manitoba
  - Isotechnika Investigational Site, Moncton, New Brunswick
  - Isotechnika Investigational Site, St. John's, Newfoundland and Labrador
  - Isotechnika Investigational Site, Halifax, Nova Scotia
  - Isotechnika Investigational Site, Hamilton, Ontario
  - Isotechnika Investigational Site, London, Ontario
  - Isotechnika Investigational Site, Maple, Ontario
  - Isotechnika Investigational Site, Markham, Ontario
  - Isotechnika Investigational Site, Newmarket, Ontario
  - Isotechnika Investigational Site, North Bay, Ontario
  - Isotechnika Investigational Site, Oakville, Ontario
  - Isotechnika Investigational Site, Oshawa, Ontario
  - Isotechnika Investigational Site, Toronto, Ontario
  - Isotechnika Investigational Site, Waterloo, Ontario
  - Isotechnika Investigational Site, Windsor, Ontario
  - Isotechnika Investigational Site, Laval, Quebec
  - Isotechnika Investigational Site, Montreal, Quebec
  - Isotechnika Investigational Site, Pointe-Claire, Quebec
  - Isotechnika Investigational Site, Sherbrooke, Quebec
  - Isotechnika Investigational Site, Ste. Foy, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gregory CR, Kyles AE, Bernsteen L, Wagner GS, Tarantal AF, Christe KL, Brignolo L, Spinner A, Griffey SM, Paniagua RT, Hubble RW, Borie DC, Morris RE. Compared with cyclosporine, ISATX247 significantly prolongs renal-allograft survival in a nonhuman primate model. Transplantation. 2004 Sep 15;78(5):681-5. doi: 10.1097/01.tp.0000131950.75697.71. PMID 15371668
- [Background] Stalder M, Birsan T, Hubble RW, Paniagua RT, Morris RE. In vivo evaluation of the novel calcineurin inhibitor ISATX247 in non-human primates. J Heart Lung Transplant. 2003 Dec;22(12):1343-52. doi: 10.1016/s1053-2498(03)00033-0. PMID 14672749
- [Background] Abel MD, Aspeslet LJ, Freitag DG, Naicker S, Trepanier DJ, Kneteman NM, Foster RT, Yatscoff RW. ISATX247: a novel calcineurin inhibitor. J Heart Lung Transplant. 2001 Feb;20(2):161. doi: 10.1016/s1053-2498(00)00290-4. No abstract available. PMID 11250240
- [Derived] Papp K, Bissonnette R, Rosoph L, Wasel N, Lynde CW, Searles G, Shear NH, Huizinga RB, Maksymowych WP. Efficacy of ISA247 in plaque psoriasis: a randomised, multicentre, double-blind, placebo-controlled phase III study. Lancet. 2008 Apr 19;371(9621):1337-42. doi: 10.1016/S0140-6736(08)60593-0. PMID 18424323

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo 1: Placebo: Placebo
- ISA247 2: voclosporin: voclosporin 0.2 mg/kg po BID
- ISA247 3: voclosporin: voclosporin: 0.3 mg/kg po BID
- ISA247 4: voclosporin: voclosporin: 0.4 mg/kg po BID
Period: Overall Study
Arm/Group | Placebo 1 | ISA247 2 | ISA247 3 | ISA247 4
Started | 115 | 107 | 113 | 116
Completed | 92 | 76 | 91 | 83
Not Completed | 23 | 31 | 22 | 33

BASELINE CHARACTERISTICS:
Groups:
- Voclosporin: 0.2: voclosporin 0.2 mg/kg po BID
- Voclosporin: 0.3: voclosporin 0.3 mg/kg po BID
- Voclosporin: 0.4: voclosporin 0.4 mg/kg po BID
- Total: Total of all reporting groups
Arm/Group | Placebo | Voclosporin: 0.2 | Voclosporin: 0.3 | Voclosporin: 0.4 | Total
Number analyzed (Participants) | 115 | 107 | 113 | 116 | 451
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 115 | 107 | 113 | 116 | 451
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 41 [19 to 63] | 42 [18 to 62] | 40 [18 to 65] | 41 [18 to 65] | 41 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 44 | 25 | 35 | 149
  Male | 70 | 63 | 88 | 81 | 302
Region of Enrollment [Number; unit: participants]
  Canada | 115 | 107 | 113 | 116 | 451

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving a PASI-75 at 12 Weeks at Each of the 3 Dose Levels of Voclosporin.
Description: Proportion of subjects achieving a PASI-75 at 12 weeks at each of the 3 dose levels of voclosporin.
Time Frame: Twelve Weeks
Measure: Count of Participants; unit: Participants
Groups:
- Voclosporin 0.2: voclosporin: voclosporin 0.2 mg/kg po BID
- Voclosporin 0.3: voclosporin: voclosporin 0.3 mg/kg po BID
- Voclosporin 0.4: voclosporin: voclosporin 0.4 mg/kg po BID
Arm/Group | Placebo | Voclosporin 0.2 | Voclosporin 0.3 | Voclosporin 0.4
Number analyzed (Participants) | 113 | 105 | 111 | 113
Participants | 4 | 14 | 26 | 44

2. Secondary Outcome: To Investigate the Safety and Tolerability of Voclosporin.
Time Frame: Twelve and twenty four weeks
Reporting Status: Not Posted

3. Secondary Outcome: To Investigate the Pharmacokinetics and Pharmacodynamics of Voclosporin After Chronic Dosing in a Subset of Subjects.
Time Frame: Twelve and twenty four weeks
Reporting Status: Not Posted

4. Secondary Outcome: To Evaluate the Effect of Voclosporin on Subject Quality of Life
Time Frame: Twelve and twenty four weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo | Voclosporin 0.2 | Voclosporin 0.3 | Voclosporin 0.4
All-Cause Mortality (participants affected / at risk) | 1/115 | 0/107 | 1/113 | 0/116
Serious Adverse Events (participants affected / at risk) | 4/115 | 2/107 | 4/113 | 1/116
Other Adverse Events (participants affected / at risk) | 62/115 | 67/107 | 65/113 | 80/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=115) | Voclosporin 0.2 (N=107) | Voclosporin 0.3 (N=113) | Voclosporin 0.4 (N=116)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parapharyngeal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct cancer (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=115) | Voclosporin 0.2 (N=107) | Voclosporin 0.3 (N=113) | Voclosporin 0.4 (N=116)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4) | 12 (14)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2) | 7 (8)
Blood pressure increased (Vascular disorders) | 5 (7) | 4 (4) | 5 (6) | 7 (7)
Glomerular Filtration Rate Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 2 (2) | 3 (3) | 11 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 6 (6) | 7 (8)
Headache (Nervous system disorders) | 12 (20) | 18 (22) | 12 (17) | 26 (34)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 27 (32) | 27 (33) | 34 (41) | 26 (32)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 12 (14) | 13 (16) | 12 (13)
Hypertension (Vascular disorders) | 7 (10) | 8 (8) | 8 (8) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No